CLINICAL TRIAL: NCT06959017
Title: Is Thromboprotection Preserved in Elderly Ostopenic Patients Who Are Severly Immobilized Before Hip Fracture?
Brief Title: Diffrence in Thromboprofilaksis in Elderly Ostoepenic Hip Fractures According to Mobility Status by Genetic Analysis
Acronym: HSP 47
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, İsmail Demirkale, Prof. Dr. İsmail Demirkale, Saglik Bilimleri Universitesi
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 01.04.2024-65
Record Dates: First submitted 2025-04-18; First posted 2025-05-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Hip Fracture of Intertrochanteric Type; Thromboembolic Event; Osteopenia; Thrombosis Embolism
Keywords: hip fracture; serpinh1; thromboembolism; rock1
MeSH Terms: conditions — Thromboembolism; Bone Diseases, Metabolic; Embolism and Thrombosis; Hip Fractures; Hereditary Sensory and Autonomic Neuropathies | interventions — Gene Expression Profiling

STUDY DESIGN:
Intervention Model Description: All patients undergo genetic expression analysis of HSP 47 (SERPİNH1, ROCK1) and the also classified by their mobility score before fracture. There is also a control group consist of age appropied healty adults
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sedentary (Active Comparator): This group is consist of the patients with pre-fracture mobility score 3-4-5
  Interventions: Genetic: Gene Expression Analysis
- Active (Experimental): This group is consist of the patients with pre-fracture mobility score 1-2
  Interventions: Genetic: Gene Expression Analysis
- Control (Experimental): This group is consist of the volunteered healty people which >65 years of age
  Interventions: Genetic: Gene Expression Analysis

INTERVENTIONS:
Genetic: Gene Expression Analysis — Each subject analysed for SERPİNH1 and ROCK1 gene exppression

SUMMARY:
Hip fracture is a common and severe disease in elderly patients. The question of the study is whether elderly patients with severe osteopenia have significantly lower levels of the collagen-binding protein Hsp47 than relatively mobile patients due to advanced immobility before the fracture, and whether they participants have a similar risk of VTE to the normal population despite having had a hip fracture and surgery.

DETAILED DESCRIPTION:
In this study, the investigators aimed to prospectively measure the Hsp 47 gene expression levels in patients scheduled for surgery due to intertrochanteric femur fracture and healthy volunteers in the same age group and compare the results with the literature.

Also the complications prior or after surgery will be compared.

ELIGIBILITY:
Inclusion Criteria:

* >65 years of age
* Interthrocanteric femur fracture AO Type 31A1, 31A2, 31A3
* Patients treated proksimal femoral nail
* Minor trauma
* Fracture mobility score 1,2,3,4,5
* Inial thrombocytes count 150.000-450.000 /µL

Exclusion Criteria:

* Body mass index >40
* Fracture mobility score 6 (unknown type)
* stage 4 chronic kidney disease
* Patients with rheumatological diseases
* Patients at serious risk of VTE(Venous thromboembolism) (according to the International Society on Thrombosis and Hemostasis, categorization of venous thromboembolism) :
* Active Hematologic Cancer
* Antiphospholipid syndrome
* History of recurrent thrombosis (DVT)
* Paroxysmal nocturnal hemoglobinuria

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
HSP 47 | Gene expression analysis will be performed once samples are collected from all participants.
  HSP 47 (SERPİNH1, ROCK1) gene expression analysis

SECONDARY OUTCOMES:
Thromboembolie | from fracture occur up to one year
  Thromboembolic events

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Demirkale, Prof Dr, Study Chair — Saglik Bilimleri Universty
Locations (1):
- Prof Dr emil Tascıoglu City Hospital, Istanbul, Şişli, Turkey (Türkiye)

REFERENCES:
- [Background] Thienel M, Muller-Reif JB, Zhang Z, Ehreiser V, Huth J, Shchurovska K, Kilani B, Schweizer L, Geyer PE, Zwiebel M, Novotny J, Lusebrink E, Little G, Orban M, Nicolai L, El Nemr S, Titova A, Spannagl M, Kindberg J, Evans AL, Mach O, Vogel M, Tiedt S, Ormanns S, Kessler B, Dueck A, Friebe A, Jorgensen PG, Majzoub-Altweck M, Blutke A, Polzin A, Stark K, Kaab S, Maier D, Gibbins JM, Limper U, Frobert O, Mann M, Massberg S, Petzold T. Immobility-associated thromboprotection is conserved across mammalian species from bear to human. Science. 2023 Apr 14;380(6641):178-187. doi: 10.1126/science.abo5044. Epub 2023 Apr 13. PMID 37053338